CLINICAL TRIAL: NCT06981208
Title: ChatGPT & Surgeon Synergy: Redefining Breast Reconstruction Consultations for Enhanced Patient Engagement and Satisfaction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 202505097
Record Dates: First submitted 2025-05-12; First posted 2025-05-20 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer; Cancer of the Breast
Keywords: Patient education; ChatGPT; Breast reconstruction
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: The surgeons will be blinded to the patient's randomization arm prior to the in-person consultation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ChatGPT-generated patient education (Experimental): * Pre-consultation ChatGPT patient education: The patients randomized into the ChatGPT education group will receive a ChatGPT patient education on paper prior to their consultation. The ChatGPT will write a patient-tailored education regarding possible reconstruction options. The patient will review this independently, without additional input or guidance from a research team member
  * Patient post-consultation survey: All patients will receive a survey after the planned in-person consultation with the plastic surgeon.
  Interventions: Other: ChatGPT-generated patient education
- Usual education (Active Comparator): - Patients will not receive any additional information prior to their consultation.
  Interventions: Other: Usual patient education
- Surgeons (No Intervention): * In order for the surgeon to be blinded to the study arm, all participants will have ChatGPT education created. Participating surgeons will review each patient education sheet prior to the consult and score the accuracy of the provided education sheet. The surgeon will proceed with the consultation as planned. The surgeon is blinded to the patient's study arm as they will be reviewing ChatGPT education for all patients. If any inaccuracies are identified in the patient education sheet, the surgeon will address this with the study team and have the errors fixed prior to providing to the patient.
  * The surgeon will receive a survey after each in-person consultation, covering patient experience, surgeon experience, and education material accuracy.

INTERVENTIONS:
Other: ChatGPT-generated patient education — This is created by entering the patient's age, medical history, social history, and case-specific details into Washington University ChatGPT Beta (HIPAA and FERPA compliant) by a study team member.
  Arms: ChatGPT-generated patient education
Other: Usual patient education — Usual patient education will include description of breast reconstruction options, with further elaboration on which option are more suitable to the patient. This include also review of risk of complications and expected recovery after surgery.
  Arms: Usual education

SUMMARY:
In this study, patients who are scheduled for breast reconstruction consultation will be randomized into the intervention group (ChatGPT-generated patient education regarding possible reconstruction options) or the control group (usual patient education). All patients will complete a survey following their in-person consultation to assess their experience and overall satisfaction with the consultation process. Additionally, participating surgeons will complete a separate survey to evaluate their consultation experience, satisfaction, and to assess the accuracy and clinical utility of the ChatGPT-generated patient education materials. The surveys are designed to gather information on patient characteristics, organizational health literacy according to Brega et al. Other survey questions have been designed to meet the outcomes of this study and have not been based on previously published surveys.

ELIGIBILITY:
Patient Eligibility Criteria:

* Scheduled for initial preoperative breast reconstruction consultation following therapeutic or prophylactic mastectomy with a surgeon at Washington University School of Medicine.
* At least 18 years of age.
* Can speak and understand English.

Surgeon Eligibility Criteria:

* Routinely performs breast reconstruction surgery at Washington University School of Medicine.
* At least 18 years of age.
* Can speak and understand English.
* Surgeon must not be a resident or fellow at time of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Estimated)
Dates: Start 2025-06-03 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Patient perceived understanding of breast reconstruction | Pre-surgical consultation (day 1)
  The patient will choose an answer ranging from 0-100 (strongly disagree to strongly agree). The higher the score, the more perceived understanding the patient had.

SECONDARY OUTCOMES:
Patient satisfaction with education regarding breast reconstruction | Pre-surgical consultation (day 1)
  The patient will choose an answer ranging from 0-100 (strongly disagree to strongly agree). The higher the score, the more satisfied the patient was.
Surgeon satisfaction with the consultation process | Pre-surgical consultation (day 1)
  Survey includes two question regarding surgeon's satisfaction with the consultation process. The surgeon will choose an answer ranging from 0-100 (strongly disagree to strongly agree). The higher the score, the more satisfied the surgeon was with the consultation process.
Surgeon perception of patient preparedness | Pre-surgical consultation (day 1)
  Survey includes one question regarding patient preparedness. The surgeon will choose an answer ranging from 0-100 (strongly disagree to strongly agree). The higher the score, the more prepared the surgeon felt the patient was.
Surgeon views on the efficiency of the consultation | Pre-surgical consultation (day 1)
  Survey includes one question regarding efficiency of the consultation. The surgeon will choose an answer ranging from 0-100 (strongly disagree to strongly agree). The higher the score, the more efficient the surgeon felt the consult was.
Surgeon overall experience with the consultation | Pre-surgical consultation (day 1)
  Survey includes one question regarding the pre-surgical consultation overall experience. The surgeon will choose an answer ranging from 0-100 (strongly disagree to strongly agree). The higher the score, the better the overall experience was.

CONTACTS AND LOCATIONS:
Overall Officials: Saif M Badran, M.D., Ph.D., FRCS, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu